CLINICAL TRIAL: NCT07043426
Title: THRIVE-DM: Improving Diabetes Care With Strategies For Addressing Health-Related Social Needs and Community Partnerships
Brief Title: Improving Diabetes Care With Strategies For Addressing Health-Related Social Needs and Community Partnerships
Acronym: THRIVE-DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-45851; 1R01DK140570-01 (NIH)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: THRIVE-DM; Community-based organizations; Triage
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Eligible participants will be categorized into low social services need (Low-SS) and high social services need (High-SS) and then randomized into intervention or control arms using block randomization in REDCap.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention- THRIVE-DM (Experimental): Participants randomized to the intervention group will receive care through the enhanced THRIVE-DM model. A Community Health Worker (CHW) will utilize the triage tool - an EPIC based tool- an EPIC based tool that categorizes patients into Low-SS or High-SS classifications based on their HRSN complexity and self-efficacy proxies.
  Interventions: Other: THRIVE-DM
- Control- Standard of care (Active Comparator): Participants randomized to the control group will be evaluated under an intention-to-treat framework. These participants will continue to receive routine clinical care.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: THRIVE-DM — Low-SS and High-SS will be referred by the CHW to appropriate community-based organizations through the THRIVE Directory. High-SS participants will also receive additional support from a patient navigator (PN), who will follow up to facilitate service connection and address barriers to engagement. CHWs and PNs will coordinate care to ensure services are aligned with the patient's assessed needs.
  Arms: Intervention- THRIVE-DM
Other: Standard of care — Standard of care may include support from the primary care team, health related social needs (HRSN) screening via the THRIVE screener, printed resource guides, and referrals to community-based organizations initiated at the discretion of clinic staff using the THRIVE Directory.
  Arms: Control- Standard of care

SUMMARY:
The goal of this study is to develop, implement, and evaluate a patient-centered triage and referral model designed to improve health outcomes for individuals with uncontrolled type 2 diabetes mellitus (T2DM) and unmet health-related social needs. The intervention builds on the existing THRIVE infrastructure at Boston Medical Center (BMC), which includes screening for social needs and a resource referral guide. It integrates medical and social care by embedding a data-driven triage tool within the EPIC electronic health record system, engaging community health workers trained in population health, and initiating closed-loop EPIC integrated referrals to community-based organizations.

This study will use a hybrid type 3 effectiveness-implementation trial design to evaluate the implementation of the THRIVE-DM intervention at the clinic level. Preliminary effectiveness will be assessed by comparing THRIVE-DM to usual care in its ability to increase patient connections to community-based organizations and improve clinical outcomes. Using a stratified randomization approach, the investigators will compare referral closure rates, receipt of social services, hemoglobin A1C levels, and patterns of health service utilization between patients enrolled in THRIVE-DM and those receiving standard care

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Must have a diagnosis of Type 2 Diabetes Mellitus (T2DM), confirmed by a current diagnosis in the medical record or at least two billing codes in the last two years, or an HbA1c level ≥6.5% in the last two years.
* Uncontrolled T2DM: Must have an HbA1c ≥9% at the time of screening.
* Health-Related Social Needs: Must have been screened for health related social needs (HRSNs) during a General Internal Medicine (GIM) visit in the last 3 months and screened positive for at least one HRSN.

Exclusion Criteria:

* Patients enrolled in Complex Care Management (CCM).
* Patients receiving hospice care.
* Patients who are deceased
* Patients with Type 1 Diabetes Mellitus (T1DM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants that connect to Community-Based Organizations | 3 months, 6 months, 3 months post intervention
  Connection to Community-Based Organizations will be assessed through several sources and documented in REDCap
Number of participants that are helped by Community-Based Organizations | 3 months, 6 months, 12 months post intervention
  Data will be collected from participant interviews
Changes in HbA1c | 3 months, 6 months, 12 months post intervention
  HbA1c data will be extracted from the EPIC electronic health record (EHR).

SECONDARY OUTCOMES:
Number of participants hospitalized | 3 months, 6 months, 12 months post intervention
  Data will be obtained from the EHR.
Number of participants that had an emergency department visit | 3 months, 6 months, 12 months post intervention
  Data will be obtained from the EHR.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fischer, MD, Principal Investigator — Boston Medical Center, Internal Medicine
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No